CLINICAL TRIAL: NCT05455983
Title: Relationship Between Different Types of COVID-19 Vaccine and Development of Immune Thrombocytopenic Purpura
Brief Title: COVID-19 Vaccine and Development of Immune Thrombocytopenic Purpura
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shymaa Mohamed Ismail, doctor, Assiut University
Other Study IDs: COVID-19 and ITP
Record Dates: First submitted 2022-07-12; First posted 2022-07-13 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: COVID-19 Vaccine
MeSH Terms: interventions — COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: covid19 vaccines — different types of (COVID-19) vaccination

SUMMARY:
Detect development of immune thrombocytopenic purpura (ITP) after different types of (COVID-19) vaccination

DETAILED DESCRIPTION:
Immune thrombocytopenia (ITP) is an acquired hemorrhagic diathesis characterized by a platelet count of < 100×109/L caused by immune-mediated destruction of platelets, impaired production or increased splenic sequestration. Primary ITP is a hematologic disorder characterized by isolated thrombocytopenia (platelet count of <100,000/uL) without associated leukopenia or anemia , without changes of the bone marrow and representing about 80% of cases. Secondary ITP is defined as any form of ITP other than the primary kind and usually secondary to an underlying precipitating etiology, as autoimmune pathology (e.g. systemic lupus erythematosus), viral infections (chronic hepatitis C virus, HIV, CMV, or varicella-zoster virus), medications, rheumatologic disorders, lymphoproliferative neoplasms. The term of acute ITP, recently replaced by newly diagnosed ITP, has less than 3 months from diagnosis. Persistent ITP refers to immune thrombocytopenia with 3 months to 1-year evolution, whereas chronic ITP is the disease longer than 12 months. Refractory ITP comprises cases which did not respond to splenectomy or relapsed after surgery, with high risk of bleeding, which makes it necessary to continue therapy.

The pathophysiology of ITP is uncertain; however, it is theorized that the acquired thrombocytopenia results from pathologic antiplatelet antibodies, impaired megakaryocytopoiesis, and T-cell-mediated destruction of platelets. ITP is primarily a diagnosis of exclusion, and the main characteristic of the disease is an increased peripheral destruction of platelets, the majority of patients showing anti-platelet membrane glycoproteins antibodies.

Patients may be asymptomatic at presentation or they may present with mild mucocutaneous to life-threatening bleeding, the intracranial one presenting the highest risk, Mortality by hemorrhage is 5% of cases.

The recent global pandemic of coronavirus disease 2019 (COVID-19) has led to vaccination in many parts of the world for herd immunity, and as vaccination has progressed, several rare adverse events have been reported. ITP has been associated with several types of vaccinations. Vaccine-related thrombocytopenia is considered to be of immune origin because antibodies can be detected on platelets in about 79% of cases. Various reports have shown that all of the live, attenuated viruses in the measles, mumps, and rubella (MMR) vaccine can cause ITP. Past studies have shown that the risk of developing ITP also increases after the administration of hepatitis A, varicella, and diphtheria-tetanus-pertussis vaccines in children and adolescents. Recently, a few case reports have shown a temporal relationship between receiving the coronavirus disease 2019 (COVID-19) vaccine and developing ITP of varying severity.

The Vaccine Adverse Effect Reporting System (VAERS) is a passive, voluntary reporting system that collects reports of adverse events associated with vaccination. VAERS reports can be submitted voluntarily by anyone, including healthcare providers, patients, or family members. A review of VAERS data has revealed 22 reports of thrombocytopenia and 13 reports of ITP following COVID-19 vaccine administration. However, underreporting is one of the main limitations of passive surveillance systems including VAERS, and it is possible that the true number of cases is far higher, especially considering that most cases of ITP are asymptomatic.

It is impossible to strictly differentiate between vaccine-induced secondary ITP and incidental primary ITP that occurred soon after vaccination. However, of the cases identified so far, 22 occurred after the first vaccination and only one after the second vaccination. Since the frequencies of occurrence are highly uneven, there is likely to be a causal relationship between the COVID-19 vaccine and the development of ITP. Lee et al. also reported that symptoms of bleeding occurred between 1 and 23 days (median 5 days) after vaccine administration.

ELIGIBILITY:
Inclusion Criteria:

* All Persons newly received COVID-19 vaccine at assiut university hospital from Decemper 2021 to April 2023 are eligible to be targeted and included in the study

Exclusion Criteria:

1. Patients who already diagnosed ITP
2. Patients with other possible causes of thrombocytopenia
3. Patients with autoimmune disorders

Ages: 17 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All Persons newly received COVID-19 vaccine at assiut university hospital from Decemper 2021 to April 2023 are eligible to be targeted and included in the study.
  Each patient will be submitted to:
  1. complete physical examination
  2. complete blood count
  3. virulogy markers
  4. liver and kidney functions
  5. Antinuclear antibody(ANA),antibody to double stranded DNA antigen (antidsDNA) Follow up with CBC after two weeks and one month following the first and second dose of the vaccination
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
different types of COVID19 vaccines and development of ITP | Baseline
  detect development of immune thrombocytopenic purpura (ITP) after different types of (COVID-19) vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed F Thabet, Professor, Study Director — Assiut University; Rania M Hafez, Assist. Prof, Study Chair — Assiut University; Shymaa M Ismail, Doctor, Principal Investigator — Assiut University
Locations (1):
- Egypt, Asyut, Egypt

REFERENCES:
- [Result] Provan D, Arnold DM, Bussel JB, Chong BH, Cooper N, Gernsheimer T, Ghanima W, Godeau B, Gonzalez-Lopez TJ, Grainger J, Hou M, Kruse C, McDonald V, Michel M, Newland AC, Pavord S, Rodeghiero F, Scully M, Tomiyama Y, Wong RS, Zaja F, Kuter DJ. Updated international consensus report on the investigation and management of primary immune thrombocytopenia. Blood Adv. 2019 Nov 26;3(22):3780-3817. doi: 10.1182/bloodadvances.2019000812. PMID 31770441
- [Result] Kistangari G, McCrae KR. Immune thrombocytopenia. Hematol Oncol Clin North Am. 2013 Jun;27(3):495-520. doi: 10.1016/j.hoc.2013.03.001. PMID 23714309
- [Result] El Ghannam D, Fawzy IM, Azmy E, Hakim H, Eid I. Relation of interleukin-10 Promoter Polymorphisms to Adult Chronic Immune Thrombocytopenic Purpura in a Cohort of Egyptian Population. Immunol Invest. 2015;44(7):616-26. doi: 10.3109/08820139.2015.1064948. PMID 26436850
- [Result] Julian JA, Mathern DR, Fernando D. Idiopathic Thrombocytopenic Purpura and the Moderna Covid-19 Vaccine. Ann Emerg Med. 2021 Jun;77(6):654-656. doi: 10.1016/j.annemergmed.2021.02.011. Epub 2021 Feb 12. No abstract available. PMID 34030782
- [Result] Cortelazzo S, Finazzi G, Buelli M, Molteni A, Viero P, Barbui T. High risk of severe bleeding in aged patients with chronic idiopathic thrombocytopenic purpura. Blood. 1991 Jan 1;77(1):31-3. PMID 1984800
- [Result] Cecinati V, Principi N, Brescia L, Giordano P, Esposito S. Vaccine administration and the development of immune thrombocytopenic purpura in children. Hum Vaccin Immunother. 2013 May;9(5):1158-62. doi: 10.4161/hv.23601. Epub 2013 Jan 16. PMID 23324619
- [Result] Du J, Xiang Y, Sankaranarayanapillai M, Zhang M, Wang J, Si Y, Pham HA, Xu H, Chen Y, Tao C. Extracting postmarketing adverse events from safety reports in the vaccine adverse event reporting system (VAERS) using deep learning. J Am Med Inform Assoc. 2021 Jul 14;28(7):1393-1400. doi: 10.1093/jamia/ocab014. PMID 33647938